CLINICAL TRIAL: NCT01314950
Title: Alzheimer's Disease Multiple Intervention Trial
Acronym: ADMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Regenstrief Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AG034946-01A1 (NIH); R01AG034946-01A1 (NIH)
Record Dates: First submitted 2011-03-10; First posted 2011-03-15 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best practices primary care (Active Comparator): Best practices primary care encompasses the collaborative care intervention tested in a prior clinical trial (Callahan CM et al. JAMA 2006).
  Interventions: Behavioral: Best practices primary care
- Home based occupational therapy (Experimental): The intervention group receives all of the components of best practice primary care in addition to a home-based intervention designed to slow functional decline.
  Interventions: Behavioral: Home based occupational therapy

INTERVENTIONS:
Behavioral: Home based occupational therapy — An occupational therapist (OT) will deliver the home-based intervention. There are three cycles of intervention over two years, with each cycle delivering eight 60-90 minute home sessions. Cycle one takes place over 16 weeks, cycle two over 32 weeks, and cycle three over one year. Telephone calls take place in intervening weeks, with additional phone calls allowed to assist with problem solving and interval problems. At minimum, the OT will perform an assessment at the beginning of each cycle in order to tailor the home based component for individual dyads at each cycle. The OT will collaborate with the patients and caregivers to develop client centered goals with "homework" each week in order to encourage carryover of strategies, home environmental modifications, or home exercise programs.
  Arms: Home based occupational therapy
Behavioral: Best practices primary care — Collaborative care is provided by an advanced practice nurse working in collaborations with a family caregiver, the primary care physician, and geriatric medicine specialists. Caregivers complete a formal assessment of problematic behaviors to assess current symptoms and stressors, and the care manager makes recommendations based on these results and using standardized protocols. Protocols focus first on non-pharmacologic interventions. If these interventions fail, the care manager collaborates with the primary care physician and/or specialists to institute protocol-based drug therapy or other strategies. Patients and caregivers are also offered access to support groups.
  Arms: Best practices primary care

SUMMARY:
The purpose of this study is to conduct a two-year randomized, controlled clinical trial to improve functioning among older adults with Alzheimer's disease by comparing a control group receiving best practices primary care with an intervention group receiving best practice primary care plus a home-based occupational therapy intervention.

DETAILED DESCRIPTION:
The proposed study builds on our findings from a previous clinical trial that demonstrated the effectiveness of collaborative care for older adults with Alzheimer's disease cared for in primary care practices. In the prior trial, we demonstrated that guideline-level medical care resulted in improved quality of care and improved behavioral and psychological symptoms over one year among patients and their caregivers. However, despite finding significant differences among study groups on Neuropsychiatric Inventory scores, we did not find a significant difference between groups in functional decline. Both study groups experienced a significant decline in function over 18 months. The current study proposes to test a home-based intervention specifically designed to slow the rate of functional decline among older adults with Alzheimer's disease.

In addition to building on our past research, the study also builds from recently reported research which demonstrated the short-term efficacy of home-based occupational therapy interventions among older adults with dementia. These trials show that older adults with dementia, including Alzheimer's disease, can both participate in and benefit from occupational therapy-based interventions delivered in the home.

The specific aim of this study is to conduct a two-year, randomized, controlled clinical trial to improve functioning among older adults with Alzheimer's disease by comparing a control group receiving best practices primary care with an intervention group receiving best practice primary care plus a home-based occupational therapy intervention. We will test the primary hypothesis that subjects with Alzheimer's disease in the intervention group will have improved function at two years compared with the best practice primary care control group.

ELIGIBILITY:
Patient Inclusion Criteria:

* Currently a patient within Wishard Health Services in Central Indiana
* Diagnosed with possible or probable Alzheimer's Disease
* Age 45 or older
* English speaking
* Hear well enough to answer questions in person or by telephone
* Community-dwelling (includes senior communities, but not skilled nursing facilities)
* Caregiver willing to participate in the study
* Willing to receive home visits
* Lives in Indianapolis metro area and planning to continue care at primary care clinic

Caregiver Inclusion Criteria

* Age 18 or older
* English speaking
* Hear well enough to answer questions in person or by telephone
* Community-dwelling
* Willing to receive home visits

Exclusion Criteria:

* Not a current patient within Wishard Health Services
* Does not speak English
* Currently enrolled in another study
* Non-community dwelling, or residing in a skilled nursing facility

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS - ADLI) | 24 months

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, 6 months, 12 months, 18 months, and 24 months
  Includes Side by Side Stand, Semi-Tandem Stand, Tandem Stand, Repeated Chair Stands, and 3 or 4 meter walk
Tandem Stand, eyes closed | Baseline, 6 months, 12 months, 18 months, and 24 months
One Leg Stand, eyes open | Baseline, 6 months, 12 months, 18 months, and 24 months
Mini Mental State Examination | Baseline, 6 months, 12 months, 18 months, and 24 months
Word List Learning | Baseline, 6 months, 12 months, 18 months, and 24 months
Delayed Word List Recall | Baseline, 6 months, 12 months, 18 months, and 24 months
Grip Strength | Baseline, 6 months, 12 months, 18 months, and 24 months
Neuropsychiatric Inventory (NPI) | Baseline, 6 months, 12 months, 18 months, and 24 months
Alzheimer's Disease Cooperative Studies Resource Use Scale | Baseline, 6 months, 12 months, 18 months, and 24 months
PHQ - 9 | Baseline, 6 months, 12 months, 18 months, and 24 months
  Depression
GAD - 7 | Baseline, 6 months, 12 months, 18 months, and 24 months
  Anxiety
Comorbid Conditions | Baseline, 6 months, 12 months, 18 months, and 24 months
Adverse Events | Baseline, 6 months, 12 months, 18 months, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Callahan, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Wishard Health Services, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Callahan CM, Boustani MA, Unverzagt FW, Austrom MG, Damush TM, Perkins AJ, Fultz BA, Hui SL, Counsell SR, Hendrie HC. Effectiveness of collaborative care for older adults with Alzheimer disease in primary care: a randomized controlled trial. JAMA. 2006 May 10;295(18):2148-57. doi: 10.1001/jama.295.18.2148. PMID 16684985
- [Background] Callahan CM, Boustani M, Sachs GA, Hendrie HC. Integrating care for older adults with cognitive impairment. Curr Alzheimer Res. 2009 Aug;6(4):368-74. doi: 10.2174/156720509788929228. PMID 19689236
- [Background] Guerriero Austrom M, Damush TM, Hartwell CW, Perkins T, Unverzagt F, Boustani M, Hendrie HC, Callahan CM. Development and implementation of nonpharmacologic protocols for the management of patients with Alzheimer's disease and their families in a multiracial primary care setting. Gerontologist. 2004 Aug;44(4):548-53. doi: 10.1093/geront/44.4.548. PMID 15331812
- [Derived] Callahan CM, Boustani MA, Schmid AA, LaMantia MA, Austrom MG, Miller DK, Gao S, Ferguson DY, Lane KA, Hendrie HC. Targeting Functional Decline in Alzheimer Disease: A Randomized Trial. Ann Intern Med. 2017 Feb 7;166(3):164-171. doi: 10.7326/M16-0830. Epub 2016 Nov 22. PMID 27893087
- [Derived] Callahan CM, Boustani MA, Schmid AA, Austrom MG, Miller DK, Gao S, Morris CS, Vogel M, Hendrie HC. Alzheimer's disease multiple intervention trial (ADMIT): study protocol for a randomized controlled clinical trial. Trials. 2012 Jun 27;13:92. doi: 10.1186/1745-6215-13-92. PMID 22737979